CLINICAL TRIAL: NCT02066623
Title: German-Austrian Register to Evaluate the Short and Long-term Safety and Therapy Outcomes of the ABSORB Everolimus-eluting Bioresorbable Vascular Scaffold System in Patients With Coronary Artery Stenosis
Brief Title: Observational Study to Evaluate Short and Long-term Safety of the ABSORB Scaffold
Acronym: GABI-R
Status: Completed | Type: Observational
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: GABI-R
Record Dates: First submitted 2014-01-20; First posted 2014-02-19 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Stenosis
Keywords: coronary artery stenosis, vascular scaffold, ABSORB
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Implantation of ABSORB Scaffold: Patients suffering from coronary artery stenosis with an indication for implantation of ABSORB scaffold
  Interventions: Device: ABSORB Scaffold

INTERVENTIONS:
Device: ABSORB Scaffold — Implantation of a drug-eluting vascular scaffold, which is completely resorbable to improve the blood flow in coronary arteries in the presence of stenosis
  Other Names: ABSORBTM Everolimus-eluting Bioresorbable Vascular Scaffold

SUMMARY:
The German-Austrian ABSORB Register shall provide an analysis of acute and long-term safety as well as therapy outcomes of the ABSORB (trade mark) bioresorbable vascular scaffold system in patients suffering from coronary artery disease.

DETAILED DESCRIPTION:
The register collects prospective data regarding the quality of care of this therapy concept including specifically the following objectives:

* Documentation of all consecutive patients having been treated with the ABSORB biore-sorbable vascular scaffold system under clinical real-world conditions
* Documentation of indications, procedural results, and short and long-term outcomes
* Documentation of the technical performance of ABSORB implant procedures
* Collection of safety data, in particular documentation of hospital mortality, major non-fatal complications (especially myocardial infarction, Re-PCI (percutaneous coronary intervention) or CABG (coronary artery bypass grafting), stroke, thrombosis)
* Documentation of long-term patient safety marked by mortality and major non-fatal complications (especially myocardial infarction, Re-PCI or CABG, stroke, thrombosis) at 30 days, 6 months, 2 years and 5 years
* Gathering of health economics data (capture of direct costs, especially with view to change of medication and outpatient/inpatient hospital services, and indirect costs) pre and post ABSORB implant
* Gathering data on the quality of life pre and post ABSORB implant to document individual QoL dimensions as well as QALY (quality adjusted life year) data

ELIGIBILITY:
Inclusion Criteria:

* ABSORB implant scheduled
* Age 18+
* Patients giving consent to keep scheduled follow-ups
* Signed informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in Germany and Austria having been implanted with ABSORB scaffold system
Sampling Method: Probability Sample
Enrollment: 3330 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse cardiac events | 5 years after index procedure
  The following events will be evaluated:
  * Death
  * Myocardial infarction
  * Clinically motivated target vessel revascularization
  * Clinically motivated target lesion revascularization
  * Composite target parameter of the aforementioned events (MACE, major adverse cardiac event) as the primary target parameter
  * Stroke
  * Composite target parameter of the aforementioned events including stroke as the primary target parameter (MACCE, major adverse cardiac and cerebrovascular event)
  * Stent thrombosis

SECONDARY OUTCOMES:
Success of ABSORB implantation | during implantation of ABSORB scaffold
  The following parameters will be evaluated to assess procedural outcome:
  * Technical success: If the residual stenosis is less than 30% in the ABSORB covered lesion segment at the end of the procedure based on visual estimation
  * Therapy success: Technical success and no periprocedural complications
  * Clinical success: Therapy success and no serious adverse cardiac (and cerebrovascular) events (MACE, MACCE)
  * TIMI (thrombolysis in myocardial infarction) flow pre and post implant
  * Sudden occlusion of side branch in the case of bifurcation stenosis
  * Optional: Quantitative coronary angiography (QCA) with index treatment: final in-scaffold and in-segment percentage diameter stenosis (%DS), reference vessel diameter

OTHER OUTCOMES:
Effectiveness of ABSORB implantation | 5 years follow-up period
  Effectiveness of ABSORB implantation will be assessed based on the following parameters:
  * Target vessel failure (TVF): This includes cardiac death, target vessel myocardial infarction (Q-wave or non-Q-wave MI) or clinically motivated target vessel revascularization (TVR), percutaneous or surgical.
  * Target lesion failure (TLF): This includes cardiac death, target vessel myocardial infarction (Q-wave or non-Q-wave MI) or clinically motivated target lesion revascularization (TLR), percutaneous or surgical.
Change in quality of life | 5 years follow-up period
  Changes in quality of life will be assessed by measuring
  * Angina pectoris scores (incl. CCS score, Canadian Cardiovascular Society score) and heart failure scores (NYHA, New York Heart Association score)
  * Standardized questionnaire for quality of life (EQ-5D)
  * Standardized questionnaire for health-related quality of life of patients with coronary artery disease (Seattle Angina Questionnaire, SAQ)
Health-economical effects of ABSORB scaffold implantation | 5 years follow-up period
  Health-economical effects will be assessed by measuring
  * Direct costs: medication, visits to general practitioners and specialists, hospitalizations, inpatient and outpatient rehab, patient care services
  * Indirect costs: disability, reduced earning capacity

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hamm, Prof. Dr., Principal Investigator — University Clinic Giessen and Kerckhoff-Clinic Bad Nauheim
Locations (81):
- Austria (6):
  - Medizinische Universität Wien, Vienna, Vienna
  - Landeskrankenhaus-Univ.Klinikum Graz, Graz
  - LKH Graz-West, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - A.ö. Krankenhaus der Stadt Linz, Linz
  - LKH Villach, Villach
- Germany (75):
  - Ilm-Kreis-Kliniken, Arnstadt-Ilmenau, Arnstadt
  - Zentralklinik Bad Berka, Bad Berka
  - SLK-Kliniken, Klinikum am Plattenwald, Bad Friedrichshall
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Hufeland Klinikum, Bad Langensalza
  - Kerckhoff-Klinik, Bad Nauheim
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Segeberger Kliniken, Bad Segeberg
  - Caritas-Klinik Pankow, Berlin
  - Charité - Universitätsmedizin Berlin - Campus Virchow-Klinikum, Berlin
  - Charité - Universitätsmedizin Berlin-Campus Benjamin Franklin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Vivantes-Klinikum Am Urban, Berlin
  - Vivantesklinik im Friedrichshain, Berlin
  - Immanuel Klinikum Bernau, Bernau
  - Gesundheitszentrum Bitterfeld-Wolfen, Bitterfeld-Wolfen
  - St. Josef- und Elisabeth- Hospital, Bochum
  - Klinikum Links der Weser, Bremen
  - Krankenhaus Buchholz, Buchholz
  - Klinikum Coburg, Coburg
  - Herzzentrum Universitätsklinikum Köln, Cologne
  - Sana-Herzzentrum Cottbus, Cottbus
  - Kardiovaskuläres Zentrum Darmstadt, Darmstadt
  - Praxisklinik Herz und Gefässe Dresden, Dresden
  - Werner-Forßmann-Krankenhaus, Eberswalde
  - Kliniken Im Naturpark Altmühltal, Klinik Eichstätt, Eichstätt
  - Universitätsklinikum Erlangen, Erlangen
  - Alfried Krupp v. Bohlen Krankenhaus, Essen
  - Elisabeth Krankenhaus Essen, Essen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Fulda, Fulda
  - Main-Kinzig-Kliniken, Gelnhausen
  - Universitätsklinikum Gießen, Giessen
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsklinikum Greifswald, Greifswald
  - Asklepios Klinik Harburg, Hamburg
  - Asklepios Klinik St. Georg, Hamburg
  - Universitäres Herzzentrum Eppendorf, Hamburg
  - Med. Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn, Heilbronn
  - Oberhavel Kliniken-Klinik Hennigsdorf, Hennigsdorf
  - Krankenhaus Herford, Herford
  - Herz- und Gefäßzentrum Oberallgäu-Kempten, Immenstadt im Allgäu
  - Klinikum Itzehoe, Itzehoe
  - Herz- und Gefäßzentrum Oberallgäu/Kempten, Kempten
  - Stiftungsklinikum Mittelrhein, Koblenz
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Ludwigshafen, Ludwigshafen am Rhein
  - Universitätsklinikum Schleswig Holstein, Lübeck
  - Klinikum Lüdenscheid, Lüdenscheid
  - St. Marien-Hospital, Lünen
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsklinikum Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Marburg, Marburg
  - Krankenhaus St. Franziskus Mönchengladbach, Mönchengladbach
  - Deutsches Herzzentrum München, Munich
  - Isar Herz Zentrum München, Munich
  - Klinikum der Universität München , Campus Großhadern, Munich
  - Klinikum München-Bogenhausen, Munich
  - Städtisches Klinikum München - Neuperlach, Munich
  - Evangelisches Krankenhaus Mülheim, Mülheim
  - Universitätsmedizin Rostock, Rostock
  - GPR Klinikum Rüsselsheim, Rüsselsheim am Main
  - St. Marien-Krankenhaus, Siegen
  - Elbe Klinikum Stade, Stade
  - SRH Zentralklinikum Suhl, Suhl
  - Universitätsklinikum Ulm, Ulm
  - St. Marienhospital, Vechta
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - Rems-Murr-Klinik Winnenden, Winnenden
  - Heinrich-Braun-Krankenhaus, Zwickau

REFERENCES:
- [Background] Nef H, Wiebe J, Achenbach S, Munzel T, Naber C, Richardt G, Mehilli J, Wohrle J, Neumann T, Biermann J, Zahn R, Kastner J, Schmermund A, Pfannebecker T, Schneider S, Limbourg T, Hamm CW. Evaluation of the short- and long-term safety and therapy outcomes of the everolimus-eluting bioresorbable vascular scaffold system in patients with coronary artery stenosis: Rationale and design of the German-Austrian ABSORB RegIstRy (GABI-R). Cardiovasc Revasc Med. 2016 Jan-Feb;17(1):34-7. doi: 10.1016/j.carrev.2015.09.002. Epub 2015 Sep 10. PMID 26431767
- [Result] Mehilli J, Achenbach S, Woehrle J, Baquet M, Riemer T, Muenzel T, Nef H, Naber C, Richardt G, Zahn R, Gori T, Neumann T, Kastner J, Schmermund A, Hamm C. Clinical restenosis and its predictors after implantation of everolimus-eluting bioresorbable vascular scaffolds: results from GABI-R. EuroIntervention. 2017 Dec 20;13(11):1319-1326. doi: 10.4244/EIJ-D-17-00291. PMID 28649953
- [Result] Nef HM, Wiebe J, Kastner J, Mehilli J, Muenzel T, Naber C, Neumann T, Richardt G, Schmermund A, Woehrle J, Zahn R, Riemer T, Achenbach S, Hamm CW. Everolimus-eluting bioresorbable scaffolds in patients with coronary artery disease: results from the German-Austrian ABSORB RegIstRy (GABI-R). EuroIntervention. 2017 Dec 20;13(11):1311-1318. doi: 10.4244/EIJ-D-17-00330. PMID 28829745
- [Result] Wohrle J, Nef HM, Naber C, Achenbach S, Riemer T, Mehilli J, Munzel T, Schneider S, Markovic S, Seeger J, Rottbauer W, Pfannebecker T, Richardt G, Zahn R, Gori T, Kastner J, Schmermund A, Hamm CW; GABI-R Study Group. Predictors of early scaffold thrombosis: results from the multicenter prospective German-Austrian ABSORB RegIstRy. Coron Artery Dis. 2018 Aug;29(5):389-396. doi: 10.1097/MCA.0000000000000618. PMID 29649071
- [Result] Huseynov A, Baumann S, Nef H, Riemer T, Schneider S, Pfannenbecker T, Achenbach S, Mehilli J, Munzel T, Gori T, Wohrle J, Zahn R, Kastner J, Schmermund A, Richardt G, Hamm CW, Akin I. Comparison between treatment of "established" versus complex "off-label" coronary lesions with Absorb(R) bioresorbable scaffold implantation: results from the GABI-R(R) registry. Clin Res Cardiol. 2020 Mar;109(3):374-384. doi: 10.1007/s00392-019-01517-8. Epub 2019 Jun 29. PMID 31256259
- [Result] Hemetsberger R, Abdelghani M, Mankerious N, Allali A, Toelg R, Gori T, Achenbach S, Riemer T, Mehilli J, Nef HM, Naber C, Wohrle J, Zahn R, Kastner J, Schmermund A, Hamm C, Munzel T, Richardt G; GABI-R Study Group. Impact of coronary calcification on outcomes after ABSORB scaffold implantation: insights from the GABI-R registry. Coron Artery Dis. 2020 Nov;31(7):578-585. doi: 10.1097/MCA.0000000000000870. PMID 32271247
- [Result] Gori T, Achenbach S, Riemer T, Mehilli J, Nef HM, Naber C, Richardt G, Wohrle J, Zahn R, Neumann T, Kastner J, Schmermund A, Hamm C, Munzel T. Hybrid Coronary Percutaneous Treatment with Metallic Stents and Everolimus-Eluting Bioresorbable Vascular Scaffolds: 2-years Results from the GABI-R Registry. J Clin Med. 2019 May 30;8(6):767. doi: 10.3390/jcm8060767. PMID 31151213
- [Derived] Pahmeier K, Neusser S, Hamm C, Kastner J, Wohrle J, Zahn R, Achenbach S, Mehilli J, Gori T, Naber C, Nef H, Neumann T, Richardt G, Schmermund A, Claas C, Riemer T, Biermann-Stallwitz J; GABI-R Study Group. Quality of life of patients with coronary heart disease treated with the bioresorbable vascular scaffold (ABSORB): 2-year results from the GABI-R-registry. BMC Cardiovasc Disord. 2022 Aug 20;22(1):379. doi: 10.1186/s12872-022-02815-2. PMID 35987601
- [Derived] Wein B, Zaczkiewicz M, Graf M, Zimmermann O, Gori T, Nef HM, Kastner J, Mehilli J, Richardt G, Wohrle J, Achenbach S, Riemer T, Hamm C, Torzewski J. No Difference in 30-Day Outcome and Quality of Life in Transradial Versus Transfemoral Access - Results From the German Austrian ABSORB Registry (GABI-R). Cardiovasc Revasc Med. 2022 Jul;40:144-149. doi: 10.1016/j.carrev.2021.11.022. Epub 2021 Nov 24. PMID 34844868
- [Derived] Boeder NF, Kastner J, Mehilli J, Munzel T, Naber C, Neumann T, Richardt G, Schmermund A, Wohrle J, Zahn R, Riemer T, Achenbach S, Hamm CW, Nef HM; GABI-R Study Group. Predictors of scaffold failure and impact of optimized scaffold implantation technique on outcome: Results from the German-Austrian ABSORB RegIstRy. Catheter Cardiovasc Interv. 2021 Oct;98(4):E555-E563. doi: 10.1002/ccd.29829. Epub 2021 Jun 18. PMID 34143547
- [Derived] Zaczkiewicz M, Wein B, Graf M, Zimmermann O, Kastner J, Wohrle J, Thomas R, Hamm C, Torzewski J; GABI-R Study Group. Two year efficacy and safety of small versus large ABSORB bioresorbable vascular scaffolds of </=18 mm device length: A subgroup analysis of the German-Austrian ABSORB RegIstRy (GABI-R). Int J Cardiol Heart Vasc. 2020 Mar 20;27:100501. doi: 10.1016/j.ijcha.2020.100501. eCollection 2020 Apr. PMID 32258361